CLINICAL TRIAL: NCT07263568
Title: The Effect of the ICN Disaster Nursing Core Competency Training on Disaster Preparedness and Psychological Resilience in Nurses
Brief Title: The Impact of ICN Disaster Nursing Core Competency Training on Disaster Preparedness and Psychological Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nermin Uyurdağ (Other)
Responsible Party: Sponsor-Investigator, Nermin Uyurdağ, Principal Investigator, Dicle University
Organization: Dicle University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: E-52857131-050.04-740993
Record Dates: First submitted 2025-11-14; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Disaster Management; Nursing; Psychological Resilience
Keywords: Disaster Management; Nursing; Education

STUDY DESIGN:
Intervention Model Description: One group of nurses will receive ICN disaster nursing basic competency training, while another group of nurses will receive standard training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICN group (Experimental): 40 people who will receive ICN disaster nursing basic competency training
  Interventions: Other: ICN disaster nursing basic competency training will be provided
- ministry group (No Intervention): A group of 40 nurses who will receive standard disaster nursing training

INTERVENTIONS:
Other: ICN disaster nursing basic competency training will be provided — ICN disaster nursing core competency training differs from the standard disaster training provided to nurses working in hospitals. It aims to equip nurses with different skills in this area.
  Arms: ICN group

SUMMARY:
The purpose of this study is to determine whether the ICN disaster nursing basic competency training affects nurses' disaster preparedness and psychological resilience. The main question to be answered by the study is:

1- Does the ICN disaster nursing basic competency training have an effect on nurses' disaster preparedness and psychological resilience compared to other disaster training programs? The researchers will provide one group of nurses with ICN disaster nursing basic competency training and another group with their regular disaster training program. Both groups will complete a questionnaire measuring disaster preparedness and psychological resilience once before the training begins and twice at specified intervals after the training is completed.

Participants:

1. Will complete the surveys administered.
2. Both groups will participate in the training programs organized for them.

DETAILED DESCRIPTION:
The Nurse Competency Assessment Scale for Disaster Management and the Brief Psychological Resilience Scale, which have undergone validity and reliability studies, were used in the research.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being a nurse
* Being employed during the study.

Exclusion Criteria:

* Leaving the job halfway through
* Not being a nurse
* Not actually working during the research (being on leave, on sick leave, etc.).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
The number of participants in the experimental group who participated in the training and whose scores on the Nurses' Disaster Management Competency Assessment Scale increased. | Immediately after training, and at 4 and 12 weeks
  Nurses' Competency Assessment Scale for Disaster Management: The total scale and its sub-dimensions are evaluated based on mean scores. A mean score approaching 1 indicates that nurses are inadequate in disaster management, while a score approaching 5 indicates that nurses are competent in disaster management.
The number of participants in the experimental group who attended the training and whose Short-Term Endurance Scale scores increased. | Immediately after training, and at 4 and 12 weeks
  The Brief Resilience Scale is a 5-point Likert-type measurement tool. "I completely disagree" is scored as 1, and "I completely agree" is scored as 5. A high score on the scale indicates a high level of psychological resilience.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Siyami Ersek Chest, Heart, and Vascular Surgery Education and Research Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data and results of the study are planned to be published in an international open-access journal.
Supporting Information: CSR
Time Frame: The study will be published in open access.
Access Criteria: The study will be published in open access.
URL: https://pubmed.ncbi.nlm.nih.gov/